CLINICAL TRIAL: NCT01850745
Title: Evaluation of a multidìsciplinary Support Program in the Adherence and Efficacy of Peginterferon Alfa-2a and Ribavirin Therapy in Chronic Hepatitis C.
Brief Title: Multidisciplinary Support Program in Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: HMAR-MSP-CHC
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2013-05

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C virus infection (CHC)
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Retrospective control group. Usual treatment with peginterferon-2a and ribavirin. No multidisciplinary support program
- Validation cohort: Prospective group. Usual treatment with peginterferon-2a and ribavirin. Multidisciplinary support program.
  Interventions: Other: Multidisciplinary support program
- Pilot cohort: Prospective intervention group. Usual pharmacological treatment with peginterferon-2a and ribavirin. Multidisciplinary support program.
  Interventions: Other: Multidisciplinary support program

INTERVENTIONS:
Other: Multidisciplinary support program — Multidisciplinary support program that included counselling about relevance of adherence by hepatologist, nurse and pharmacist. Psychologist and psychiatrist support if needed.
  Groups: Pilot cohort; Validation cohort

SUMMARY:
Adherence to antiviral treatment in chronic hepatitis C (CHC) is an important factor to achieve sustained virological response (SVR). The aim of our study is to evaluate the efficacy of a multidisciplinary support program (MSP) in adherence to and efficacy of pegylated interferon alfa-2a and ribavirin compared to the conventional approach. We assessed 447 patients with CHC receiving antiviral treatment distributed into 3 groups: control group (recruited 2002-2004, n= 147), MSP-pilot group (recruited 2005-2006, n=131), and MSP-validation group (recruited 2007-2009, n=169).

DETAILED DESCRIPTION:
Adherence to antiviral treatment in chronic hepatitis C (CHC) is an important factor to achieve sustained virological response (SVR). The aim of our study is to evaluate the efficacy of a multidisciplinary support program (MSP) in adherence to and efficacy of pegylated interferon alfa-2a and ribavirin compared to the conventional approach. We assessed 447 patients with CHC receiving antiviral treatment distributed into 3 groups: control group (follow-up 2002-2004, n= 147), MSP-pilot group (follow-up 2005-2006, n=131), and MSP-validation group (follow-up 2007-2009, n=169).A cost-effectiveness analysis was performed using a Markov model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C eligible to receive antiviral treatment.

Exclusion Criteria:

* Patients who had undergone previous antiviral treatment, those with human immunodeficiency virus (HIV) or hepatitis B virus (HBV) co-infection, and individuals included in other treatment protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C virus infection (CHC)
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2003-01; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Sola, MD, Principal Investigator — Hsopital del Mar, Parc de Salut MAR
Locations (1):
- Hospital del Mar, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Validation Cohort | Pilot Cohort
Started | 147 | 169 | 131
Completed | 147 | 169 | 131
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Validation Cohort | Pilot Cohort | Total
Number analyzed (Participants) | 147 | 169 | 131 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (1) | 42 (1) | 42 (1) | 42 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 45 | 46 | 139
  Male | 99 | 124 | 85 | 308

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Treatment
Description: Adherent patients were defined as those receiving equal or more than 80% of total dose of pegylated interferon (180 microg/week) and ribavirin (1200 mg/d) during equal o more than 80% of duration treatment (48 weeks).
  Non-adherent patients were defined as those receiving less than 80% of total dose of pegylated interferon (180 microg/week) and ribavirin (1200 mg/d) during less than 80% of duration treatment (48 weeks).
Time Frame: 48 months
Measure: Number; unit: participants
Arm/Group | Control | Validation Cohort | Pilot Cohort
Number analyzed (Participants) | 147 | 169 | 131
participants | 116 | 155 | 124

2. Secondary Outcome: Efficacy of Treatment Measured by Sustained Virological Response
Description: The secondary efficacy end point was to evaluate the sustained virological response (SVR) of antiviral treatment.
  SVR was defined as undetectable hepatitis C virus viral load (<15 IU/ml) 24 weeks after treatment completion.
  Non-SVR was defined as detectable hepatitis C virus viral load (>15 IU/ml) 24 weeks after treatment completion.
Time Frame: baseline and 72 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Validation Cohort | Pilot Cohort
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/169 | 0/131
Serious Adverse Events (participants affected / at risk) | 2/147 | 2/169 | 2/131
Other Adverse Events (participants affected / at risk) | 52/147 | 14/169 | 4/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=147) | Validation Cohort (N=169) | Pilot Cohort (N=131)
Depression major (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=147) | Validation Cohort (N=169) | Pilot Cohort (N=131)
Anemia (Blood and lymphatic system disorders) | 52 (52) | 14 (14) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No